CLINICAL TRIAL: NCT03895918
Title: A Novel Parenting Skills Intervention to Improve Medication Adherence in Pediatric Cancer
Brief Title: Parenting Skills Intervention in Improving Medication Adherence in Pediatric Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: I 77618; NCI-2019-01554 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); I 77618 (Other: Roswell Park Cancer Institute)
Record Dates: First submitted 2019-03-28; First posted 2019-03-29 (Actual); Last update posted 2021-09-16 (Actual); Status verified 2021-09

CONDITIONS: Guardian; Hematologic and Lymphocytic Disorder; Malignant Neoplasm; Parent
MeSH Terms: conditions — Hematologic Diseases; Neoplasms | interventions — Remote Patient Monitoring

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Delayed Group (delayed parental skills) (Experimental): Participants continue medication adherence monitoring over 2 weeks and then receive parental skills intervention sessions consisting of 4 integrated components: creating consistent medication routines, education in child management strategies, strategies for helping children adhere to medication, and training in specific parental behavioral techniques over 30 minutes weekly for 4 weeks.
  Interventions: Other: Educational Activity; Procedure: Patient Monitoring; Other: Questionnaire Administration
- Early Group (early parental skills) (Experimental): Participants continue medication adherence monitoring over 1 week and then receive parental skills intervention sessions consisting of 4 integrated components: creating consistent medication routines, education in child management strategies, strategies for helping children adhere to medication, and training in specific parental behavioral techniques over 30 minutes weekly for 4 weeks.
  Interventions: Other: Educational Activity; Procedure: Patient Monitoring; Other: Questionnaire Administration
- Late Group (late parental skills) (Experimental): Participants continue medication adherence monitoring over 3 weeks and then receive parental skills intervention sessions consisting of 4 integrated components: creating consistent medication routines, education in child management strategies, strategies for helping children adhere to medication, and training in specific parental behavioral techniques over 30 minutes weekly for 4 weeks.
  Interventions: Other: Educational Activity; Procedure: Patient Monitoring; Other: Questionnaire Administration

INTERVENTIONS:
Other: Educational Activity — Undergo parenting skills intervention
Procedure: Patient Monitoring — Undergo medication adherence monitoring
  Other Names: monitor
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This trial studies how well a parenting skills intervention works in improving medication adherence in pediatric cancer patients. The parenting skills intervention provides support and skills training to parents who administer medicine daily to their child and may improve the childs taking of medications correctly as prescribed by the doctor. Ultimately, this may improve treatment outcomes, among children who are experiencing an illness.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To pilot test a novel parenting intervention. II. To examine the feasibility and preliminary efficacy of the parenting intervention on child medication adherence among children who are experiencing an illness.

OUTLINE: Participants with poor medication adherence are randomized to 1 of 3 groups.

EARLY GROUP: Participants continue medication adherence monitoring over 1 week and then receive parental skills intervention sessions consisting of 4 integrated components: creating consistent medication routines, education in child management strategies, strategies for helping children adhere to medication, and training in specific parental behavioral techniques over 30 minutes weekly for 4 weeks.

DELAYED GROUP: Participants continue medication adherence monitoring over 2 weeks and then receive parental skills intervention sessions consisting of 4 integrated components: creating consistent medication routines, education in child management strategies, strategies for helping children adhere to medication, and training in specific parental behavioral techniques over 30 minutes weekly for 4 weeks.

LATE GROUP: Participants continue medication adherence monitoring over 3 weeks and then receive parental skills intervention sessions consisting of 4 integrated components: creating consistent medication routines, education in child management strategies, strategies for helping children adhere to medication, and training in specific parental behavioral techniques over 30 minutes weekly for 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Be a parent of a child (2 to 10 years old) with any hematology or oncology diagnosis who is receiving treatment at Roswell Park Comprehensive Cancer Center. We define parents as biological parents, adoptive parents, foster parents, stepparents, and legal guardians
* Parent must have primary medication responsibility
* The child's treatment must include home-based daily oral medication
* Parent must have verbal English fluency
* Participant or legal representative must understand the investigational nature of this study and sign an Independent Ethics Committee/Institutional Review Board approved written informed consent form prior to receiving any study related procedure

Exclusion Criteria:

* Be a parent of a pediatric patient with any hematology or oncology diagnosis who is receiving treatment at Roswell Park and is < 2 or > 10 years old
* Parent does not have primary medication responsibility
* Child's treatment does not include home-based daily oral medication
* Parent does not have verbal English fluency
* If unable to consent or a prisoner
* Unwilling or unable to follow protocol requirements
* Any condition which in the investigator?s opinion deems the participant an unsuitable candidate to receive study intervention

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2019-01-03 (Actual); Primary Completion 2020-11-25 (Actual); Study Completion 2020-11-25 (Actual)

PRIMARY OUTCOMES:
Objective medication adherence | Up to 4 weeks post study
  Assessed using Medication Event Monitoring Systems (MEMS) track caps.The project manager will conduct reviews of each child?s medical record to obtain data on the medication dose prescribed each day and dates when the medication was held for illness or toxicity. MEMS-based adherence variables will be constructed as a percentage based upon the ratio of the number of days with MEMS cap openings (X) to the number of days the medication was prescribed (N). Will remove days when the medication was held by the prescriber from the denominator (X/N x 100).

SECONDARY OUTCOMES:
Change in parenting stress | Baseline up to 4 weeks post study
  Pre and post intervention 15minute surveys
Intervention feasibility | Up to 4 weeks post study
  Assessed using survey assessments
Change in parenting behaviors | Baseline up to 4 weeks
  Pre and Post intervention 15 minute surveys

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Bouchard, Principal Investigator — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States